CLINICAL TRIAL: NCT06270225
Title: A Randomized, Open-label, Active-Controlled Phase II Trial to Evaluate the Efficacy and Safety of SSGJ-613 for Prophylaxis Against Acute Gouty Arthritis Flares in Subjects Initiating Urate-Lowering Treatment.
Brief Title: A Study of SSGJ-613 in Gout Subjects Initiating Urate-Lowering Treatment.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-613-PGF-II-01
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Gout Arthritis
MeSH Terms: conditions — Arthritis, Gouty | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SSGJ-613 100 mg (Experimental): Subjects will receive 100mg SSGJ-613 on Day 1.
  Interventions: Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 100 mg
- SSGJ-613 200 mg (Experimental): Subjects will receive 200mg SSGJ-613 on Day 1.
  Interventions: Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 200 mg
- Colchicine 0.5mg (Active Comparator): Subjects will receive 0.5mg/d Colchicine for 12 weeks.
  Interventions: Drug: Colchicine 0.5 mg

INTERVENTIONS:
Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 100 mg — Subjects will receive one s.c. injection of SSGJ-613 on Day 1.
  Other Names: SSGJ-613 100mg
  Arms: SSGJ-613 100 mg
Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 200 mg — Subjects will receive one s.c. injection of SSGJ-613 on Day 1.
  Other Names: SSGJ-613 200mg
  Arms: SSGJ-613 200 mg
Drug: Colchicine 0.5 mg — Subjects will receive 0.5mg/d Colchicine for 12 weeks.
  Arms: Colchicine 0.5mg

SUMMARY:
The purpose of this study is to determine the efficacy and safety of recombinant anti-interleukin-1β humanized monoclonal antibody injection in Chinese gout participants Initiating Urate-Lowering Treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 Years to 75 Years, both male and female.
* BMI ≤40 kg/m2.
* Meeting the American College of Rheumatology (ACR) 2015 criteria for the classification of gouty arthritis.
* ≥2 acute gout flares within 1 year prior to screening.
* Willingness to initiate urate-lowering treatment or to initiate urate-lowering treatment within 7 days prior to administration.

Exclusion Criteria:

* Gout caused by radiotherapy/chemotherapy, organ transplantation, tumors, etc.
* Evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis.
* Presence of severe renal function impairment.
* Intolerance of subcutaneous injection.
* Known presence or suspicion of active or recurrent bacterial, fungal, or viral infection at the time of enrollment.
* Live vaccinations within 8 weeks prior to the start of the study.
* Use of forbidden therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Numbers of acute gout flares | 12 weeks

SECONDARY OUTCOMES:
Numbers of acute gout flares | 24 weeks
Proportions of subjects with at least 1 acute gout flare | 12 weeks
Proportions of subjects with at least 1 acute gout flare | 24 weeks
Time from randomization to first acute flare. | 24 weeks
Duration of acute gout flares. | 12 weeks
Duration of acute gout flares. | 24 weeks
Subject's overall assessment of response to treatment | 24 weeks
  Response to treatment will be assessed by the subjects using a five-point Likert scale: 1-very good, 2-good, 3-fair, 4-poor, and 5-very poor.
Investigator's overall assessment of response to treatment | 24 weeks
  Response to treatment will be assessed by the Investigators using a five-point Likert scale: 1-very good, 2-good, 3-fair, 4-poor, and 5-very poor.
36-item Short Form Survey (SF-36) | 24 weeks
  36-Item Short Form Survey (SF-36) will be used to assess the health and functional changes of the subjects. It comprises 36 items that measure perceived health on eight scales (i.e., physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health) with higher scores (range 0-100) reflecting better perceived health.
Adverse events (AE) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hejian Zou, MD, Principal Investigator — Shanghai Huashan Hospital Fudan University-Rheumatology; Qinghong Zhou, Study Director — Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd.
Locations (1):
- Shanghai Huashan Hospital Fudan University-Rheumatology, Shanghai, Shanghai Municipality, China